CLINICAL TRIAL: NCT00666497
Title: A Phase 2, Randomized, Open-Label Study of Azacitidine (Vidaza) vs MGCD0103 vs Azacitidine in Combination With MGCD0103 for the Treatment of Elderly Subjects With Newly Diagnosed AML or Intermediate-2 or High-Risk MDS
Brief Title: Phase 2 Study of Azacitidine (Vidaza) vs MGCD0103 vs Combination in Elderly Subjects With Newly Diagnosed Acute Myeloid Leukemia (AML) or Myelodysplastic Syndrome (MDS)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Celgene terminated its collaboration agreement with MethylGene for the development of MGCD0103. All Celgene-sponsored trials with MGCD0103 with be closed.
Sponsor: Mirati Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 103 PH GL 2007 CL003
Record Dates: First submitted 2008-04-23; First posted 2008-04-25 (Estimated); Last update posted 2015-05-08 (Estimated); Status verified 2015-04

CONDITIONS: Acute Myeloid Leukemia (AML); Myelodysplastic Syndrome (MDS)
Keywords: Acute Myeloid Leukemia; Myelodysplastic Syndrome; Azacitidine; Vidaza; MGCD0103; Histone deacetylase inhibitor; DNA methyltransferase inhibitor; Epigenetic Therapy
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Azacitidine; mocetinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A (Experimental): Azacitidine
  Interventions: Drug: Azacitidine
- B (Experimental): MGCD0103
  Interventions: Drug: MGCD0103
- C (Experimental): Azacitidine + MGCD0103
  Interventions: Drug: Azacitidine; Drug: MGCD0103

INTERVENTIONS:
Drug: Azacitidine — 75 mg/m2/day for 5 days, subcutaneous (SC) injection, Days 1 - 5 of every 28-day cycle
  Other Names: Vidaza
  Arms: A; C
Drug: MGCD0103 — 90 mg, oral (PO) administration, 3 times per week for 12 doses, 28-day cycle
  Arms: B
Drug: MGCD0103 — 90 mg, oral (PO) administration, 3 times per week for 10 doses, 28-day cycle
  Arms: C

SUMMARY:
The purpose of the study is to determine how effective azacitidine, MGCD0103, and the combination of azacitidine and MGCD0103 are in treating AML or MDS in people over 60 years of age.

DETAILED DESCRIPTION:
This randomized, 3-arm Phase 2 study will compare the safety and efficacy of single-agent azacitidine (currently 1 of 3 approved treatments for myelodysplastic syndrome [MDS]) to that of single-agent MGCD0103 and to that of combination therapy with MGCD0103 and azacitidine in elderly patients with acute myelogenous leukemia (AML) or intermediate-2 (Int-2) or high-risk MDS, for whom no standard of care exists. The goal of the study is to determine which of the 3 treatment arms are worthy of further investigation in a subsequent Phase 3 study of elderly subjects with AML or Int-2 or high-risk MDS.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written informed consent, and be willing and able to comply with all the study procedures
* Must be 60 years of age or older
* Must have a pathologic confirmation of newly diagnosed (de novo or untreated secondary) AML or newly diagnosed Int-2 or high-risk MDS (IPSS classification) according to WHO criteria
* Must have a Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* Must have adequate organ function, including total bilirubin ≤ 1.5 x upper limit of normal (ULN); AST & ALT ≤ 2.5 x ULN; and serum creatinine ≤ 2.0 x ULN.

Exclusion Criteria:

* Considered fit for intensive chemotherapy and opt to be treated with intensive chemotherapy
* Prior transplantation or any prior anticancer therapy (standard or investigational, including chemotherapy, treatment with HDAC inhibitors, or combination HDAC and azacitidine) administered to treat AML or MDS.
* Clinical evidence of central nervous system (CNS) involvement by leukemia
* A diagnosis of promyelocytic leukemia
* Previous or concurrent malignancy except adequately treated basal cell or squamous cell skin cancer; in situ carcinoma of the cervix, or other solid tumor treated curatively, and without evidence of recurrence for at least 3 years prior to study entry
* Active and uncontrolled clinically significant infection
* Known positive serology for hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCV Ab) or human immunodeficiency virus (HIV)
* Less than 4 weeks elapsed since any major surgery
* Any prior or active disease that may interfere with the procedures or evaluations to be conducted in the study

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2008-06; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Overall response rate as assessed using IWG criteria for AML and MDS | After 45, 90, 135, and 180 subjects are enrolled and evaluated for response to treatment

SECONDARY OUTCOMES:
Duration of response; Time to progression; Progression-free survival; RBC transfusion independence; Hematologic improvement; Quality of life; Safety profile; and Pharmacokinetics of azacitidine and MGCD0103 | After 45, 90, 135, and 180 subjects are enrolled and evaluated for response to treatment

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Reid, MSc, MBA, Study Director — MethylGene Inc.
Locations (8):
- MD Anderson Cancer Center, Houston, Texas, United States
- Canada (2):
  - Diamond Centre, Leukemia/BMT Program of BC, Vancouver, British Columbia
  - Jewish General Hospital, Montreal, Quebec
- United Kingdom (5):
  - University Hospital, Birmingham
  - Royal Bournemouth Hospital, Bournemouth
  - St. Bartholomews Hospital, London
  - Kings College Hospital, London
  - John Radcliffe Hospital, Oxford

REFERENCES:
- See also: The Leukemia & Lymphoma Society — http://www.leukemia-lymphoma.org/hm_lls
- See also: The Myelodysplastic Syndromes Foundation — http://www.mds-foundation.org/
- See also: Leukemia Research Foundation — http://www.leukemia-research.org/NETCOMMUNITY/Page.aspx?pid=183&srcid=-2